CLINICAL TRIAL: NCT05612425
Title: Safety Behavior Fading Versus Unhealthy Behavior Fading for Appearance Concerns: A Randomized Controlled Trial
Brief Title: Text Message Safety Behavior Fading for Appearance Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003637
Record Dates: First submitted 2022-11-04; First posted 2022-11-10 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Body Dysmorphic Disorders; Social Anxiety Disorder; Eating Disorders
Keywords: safety behaviors; intervention; text message; appearance concerns
MeSH Terms: conditions — Body Dysmorphic Disorders; Phobia, Social; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Fading (Experimental): Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed appearance-related safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day.
  Interventions: Behavioral: Safety Behavior Fading for Appearance Concerns
- Unhealthy Behavior Fading (Active Comparator): Individuals randomly assigned to the unhealthy behavior fading condition will receive instructions to decrease or eliminate unhealthy behaviors that are unrelated to appearance. They will also receive daily reminders via text message to decrease these behaviors, along with a behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each behavior over the previous day.
  Interventions: Behavioral: Unhealthy Behavior Fading

INTERVENTIONS:
Behavioral: Safety Behavior Fading for Appearance Concerns — Participants are asked to reduce or eliminate safety behaviors via text message reminders and checklists to monitor progress.
  Arms: Safety Behavior Fading
Behavioral: Unhealthy Behavior Fading — Participants are asked to reduce or eliminate unhealthy behaviors via text message reminders and checklists to monitor progress.
  Arms: Unhealthy Behavior Fading

SUMMARY:
The current study aims to explore the efficacy of a text message based safety behavior fadinig intervention compared to an unhealthy behavior fading intervention for appearance concerns.

DETAILED DESCRIPTION:
Description: Appearance-related safety behavior fading intervention procedures will follow methodology previously used in the Cougle Lab. The safety behavior fading intervention is designed to target a decrease or elimination of appearance-related safety behaviors.

Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed appearance-related safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day.

Individuals randomly assigned to the unhealthy behavior fading condition will receive instructions to decrease or eliminate unhealthy behaviors. They will also receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day.

ELIGIBILITY:
Inclusion Criteria:

* elevated appearance concerns as defined by a score of 53 or higher on the SAAS
* Being female

Exclusion Criteria:

* being male
* Score of 52 or lower on the SAAS
* Currently receiving treatment (therapy, counseling, etc.) for anxiety, depression, eating disorder, or body image/appearance concerns
* If applicable, unstable psychiatric medication usage any time over the past 4 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Social Appearance Anxiety Scale | Day 0, Day 28, Day 56
  Self-report scale that measures appearance anxiety symptoms. Scores range from 16 to 80 with higher scores indicating higher levels of appearance concerns.
Change in Eating Disorder-15 | Day 0, Day 28, Day 56
  Self-report scale that measures eating disorder symptoms. Scores range from 0 to 90 with higher scores indicating higher levels of eating pathology.
Change in Social Phobia Inventory | Day 0, Day 28, Day 56
  Self-report scale that measures social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety.
Credibility and Expectancy Questionnaire | Day 0
  Self-report scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies.
Change in Appearance Behaviors Checklist | Day 0, Day 28, Day 56
  Self-report scale used to measure frequency of engaging in appearance related safety behaviors. This scale will be used as a manipulation check.
Change in Unhealthy Behaviors Checklist | Day 0, Day 28, Day 56
  Self-report scale used to measure frequency of engaging in unhealthy behaviors. This scale will be used as a manipulation check.
Beliefs About Appearance Scale | Day 0, Day 28, Day 56
  Self-report scale for measuring appearance importance for use in clinical outcome studies. Each item is rated on a 0-4 scale with a total score range of 0-80 with higher scores indicating greater appearance importance.
UCLA Loneliness Scale-8 | Day 0, Day 28, Day 56
  Self-report scale for measuring loneliness for use in clinical outcome studies. Total scores range from 0 to 32 with higher scores indicating higher loneliness.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Day 0, Day 28, Day 56
  Self-report measure of depression symptom severity.
Assessment of ideal self | Day 0, Day 28, Day 56
  Self-report measure of appearance importance where individuals must allocate a budget of 100 to 7 different ideals including appearance, creativity, friendliness, work ethic, intelligence, humor, and income.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel TA, Cougle JR. Safety behavior reduction for appearance concerns: A randomized controlled trial of a smartphone-based intervention. J Consult Clin Psychol. 2024 Dec;92(12):788-799. doi: 10.1037/ccp0000920. Epub 2024 Oct 24. PMID 39446647